CLINICAL TRIAL: NCT03274102
Title: A Randomized, Controlled Clinical Trial to Evaluate the Safety and Immunogenicity of Concomitant Administration of EV71 Vaccine With Recombinant Hepatitis B Vaccine/Group A Meningococcal Polysaccharide Vaccine
Brief Title: Safety and Immunogenicity of Concomitant Administration of EV71 Vaccine With EPI Vaccines
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Collaborators: Guangdong Center for Disease Prevention and Control (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PRO-EV71-4003
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2018-12

CONDITIONS: Hand, Foot and Mouth Disease
Keywords: Inactivated Enterovirus Type 71 (EV71) Vaccine; Concomitant vaccination; Safety; Immunogenicity; Infant
MeSH Terms: conditions — Hand, Foot and Mouth Disease

STUDY DESIGN:
Masking Description: open-labelled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I-EV71 vaccine and EPI vaccines (Experimental): Concomitant administration of EV71 vaccine with EPI vaccines: EV71 Vaccine (intramuscular injection,0.5ml,first dose)/recombinant hepatitis B vaccine（intramuscular injection,0.5ml）on day 0 and EV71 Vaccine (injection, 0.5ml,second dose)/ Group A meningococcal polysaccharide vaccine(subcutaneous injection, 150ug) on day 30.
  Interventions: Biological: Concomitant administration of EV71 vaccine with EPI vaccines
- Group II-EPI vaccine only (Active Comparator): Single injection of EPI vaccine: recombinant hepatitis B vaccine (intramuscular injection, 0.5ml) on day 0 and Group A meningococcal polysaccharide vaccine (subcutaneous injection,150ug) on day 30.
  Interventions: Biological: Single injection of EPI vaccine
- Group III-EV71 vaccine only (Active Comparator): EV71 Vaccine only: the first and second dose of EV71 Vaccine (intramuscular injection,0.5ml) on day 0 and day 30 respectively.
  Interventions: Biological: EV71 Vaccine only

INTERVENTIONS:
Biological: Concomitant administration of EV71 vaccine with EPI vaccines — 1. The investigated EV17 vaccine was manufactured by Sinovac Biotech Co., Ltd.； the recombinant hepatitis B vaccine was manufactured by Shenzhen Kangtai Biological Products Co., Ltd; the Group A meningococcal polysaccharide vaccine was manufactured by Wuhan Institute of Biological Products Co., Ltd.
  2. The primary vaccination schedule of hepatitis B vaccine includes 3 doses with a schedule of 0,1,6 month, and subjects only receive 3rd vaccination in this study; the primary vaccination schedule of Group A meningococcal polysaccharide vaccine includes 2 doses with 3 months interval between doses, and subjects only receive 1st vaccination in this study
  Arms: Group I-EV71 vaccine and EPI vaccines
Biological: Single injection of EPI vaccine — 1. The recombinant hepatitis B vaccine was manufactured by Shenzhen Kangtai Biological Products Co., Ltd; the Group A meningococcal polysaccharide vaccine was manufactured by Wuhan Institute of Biological Products Co., Ltd.
  2. The primary vaccination schedule of hepatitis B vaccine includes 3 doses with a schedule of 0,1,6 month, and subjects only receive 3rd vaccination in this study; the primary vaccination schedule of Group A meningococcal polysaccharide vaccine includes 2 doses with 3 months interval between doses, and subjects only receive 1st vaccination in this study
  Arms: Group II-EPI vaccine only
Biological: EV71 Vaccine only — The investigated EV17 vaccine was manufactured by Sinovac Biotech Co., Ltd.
  Arms: Group III-EV71 vaccine only

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of concomitant administration of EV71 vaccine with recombinant hepatitis B vaccine/Group A meningococcal polysaccharide vaccine.

DETAILED DESCRIPTION:
This study is an open-label, single-center, randomized, comparative phase IV clinical trial. The purpose of this study is to evaluate the safety and immunogenicity of concomitant administration of EV71 vaccine manufactured by Sinovac (Beijing) Vaccine Technology Co., Ltd. with recombinant hepatitis B vaccine/Group A meningococcal polysaccharide vaccine. 780 healthy infants of 6 months old as participants are randomly assigned into three experimental groups in the ratio 1:1:1. The group I receive EV71 Vaccine (first dose)& recombinant hepatitis B vaccine on day 0 and EV71 vaccine (second dose)& Group A meningococcal polysaccharide vaccine on day 30. The group II receive recombinant hepatitis B vaccine on day 0 and Group A meningococcal polysaccharide vaccine on day 30. The group III receive the first and second dose of EV71 Vaccine on day 0 and day 30 respectively.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers aged 6 months
* Finished two doses of vaccination (0,1 month) of hepatitis B vaccine prior to study entry
* Proven legal identity
* Guardian(s) of the volunteer should be capable of understanding the written consent form, and such form should be signed before the infant being included into this study

Exclusion Criteria:

* Finished all the three doses vaccination (0,1,6 month) of hepatitis B vaccine prior to study entry
* Prior vaccination of meningococcal polysaccharide vaccine
* Prior vaccination of EV71 vaccine
* Unable to receive vaccination on both arms
* History of hand foot and mouth disease
* Previously tested HBsAg positive
* Mother of the subject had been previously tested HBsAg positive
* History of asthma; history of allergy to any vaccine or vaccine ingredient, or serious adverse reaction(s) to vaccination, such as urticaria, difficulty in breathing, angioneurotic edema, abdominal pain, etc
* Congenital malformation, developmental disorders, genetic defects
* Autoimmune disease or immunodeficiency/immunosuppressive
* Severe nervous system disease or mental illness
* Diagnosed coagulation function abnormal (e.g., coagulation factor deficiency, coagulation disorder, or platelet abnormalities) , or obvious bruising or coagulation disorders
* Any immunosuppressant, cytotoxic medicine, or inhaled corticosteroids (except corticosteroid spray for treatment of allergic rhinitis or corticosteroid treatment on surface for acute non-complicated dermatitis) within 6 month prior to study entry
* Receipt of blood product (e.g., immunoglobulin) within 3 months prior to study entry
* Receipt of any other investigational medicine(s) within 30 days prior to study entry
* Receipt of any live attenuated vaccine within 14 days prior to study entry
* Receipt of any subunit vaccine or inactivated vaccine within 7 days prior to study entry
* Acute disease or acute stage of chronic disease within 7 days prior to study entry
* Axillary temperature > 37.0 ℃
* Any other factor that suggesting the volunteer is unsuitable for this study based on the judgement of investigators

Exclusion Criteria of the Second Injection:

* Subjects with one of the following 1 to 3 conditions are forbidden to continue vaccination, while the other study steps could be carried out based on the judgement of investigator; for subjects with one of the following 4 to 5 conditions, whether to continue vaccination are determined by the investigator; for subjects with one of the following 6 to 7 conditions, vaccination may be delayed in the time window specified in the study:

  1. Any serious adverse event that has a causal relationship with the investigated vaccine (except the group II)
  2. Severe allergic reactions or hypersensitivity after vaccination (including urticaria / rash appear within 30 minutes after vaccination, except the group II )
  3. Any confirmed or suspected autoimmune disease or immunodeficiency disease (e.g., HIV infection)
  4. New chronic diseases or acute stage of chronic diseases
  5. Other reactions (including severe pain, severe swelling, severe activity limitation, persistent hyperthermia, severe headache or other systemic or local reactions) determined by the investigators
  6. Acute diseases (moderate or severe diseases with or without fever)
  7. Axillary temperature> 37.0 ℃

Ages: 6 Months to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 780 (Actual)
Dates: Start 2017-04-22 (Actual); Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
The seropositive rate of EV71 neutralizing antibody, anti-HBs and serum bactericidal antibody 1 month after 2 doses of vaccination | 30 days after 2 doses of injection
  Immunogenicity indicator

SECONDARY OUTCOMES:
Incidence of solicited local or systemic adverse events within 7 days after each dose | 7 days after each dose of injection
  Safety indicator
Incidence of unsolicited local or systemic adverse events within 30 days after each dose | 30 days after each dose of injection
  Safety indicator
Incidence of serious adverse events during the period of safety monitoring | 60 days after the first dose injection
  Safety indicator
The seroconversion rate of EV71 neutralizing antibody, anti-HBs and serum bactericidal antibody(SBA) 1 month after 2 doses of vaccination | 30 days after 2 doses of injection
  Immunogenicity indicator
EV71 neutralizing antibody GMT, anti-HBs GMC and SBA antibody GMT 1 month after 2 doses of vaccination | 30 days after 2 doses of injection
  Immunogenicity indicator

CONTACTS AND LOCATIONS:
Overall Officials: Huizhen Zheng, Principal Investigator — Guangdong Center for Disease Prevention and Control
Locations (1):
- Dongguan Municipal Center for Disease Control and Prevention, Dongguan, Guangdong, China

REFERENCES:
- [Derived] Zhang Z, Liang Z, Zeng J, Zhang J, He P, Su J, Zeng Y, Fan R, Zhao D, Ma W, Zeng G, Zhang Q, Zheng H. Immunogenicity and Safety of an Inactivated Enterovirus 71 Vaccine Administered Simultaneously With Hepatitis B Vaccine and Group A Meningococcal Polysaccharide Vaccine: A Phase 4, Open-Label, Single-Center, Randomized, Noninferiority Trial. J Infect Dis. 2019 Jul 2;220(3):392-399. doi: 10.1093/infdis/jiz129. PMID 30891604